CLINICAL TRIAL: NCT01891929
Title: Specific Cognitive Remediation for Schizophrenia (RECOS) and Sheltered Employment: a Multicentre Controlled Randomized Trial.
Brief Title: Cognitive Remediation and Sheltered Employment in Schizophrenia
Acronym: RemedRehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Sainte Anne Hospital (Paris) (Unknown); Clermont-de-l'Oise Hospital (Clermont-de-l'Oise) (Unknown); Saint-Egrève Hospital (Saint-Egrève) (Unknown); Centre Hospitalier de Niort (Other); Sainte-Marguerite Hospital (Marseille) (Unknown); Centre Hospitalier Henri Laborit (Other); University Hospital, Tours (Other); Mental Health Center MGEN (Rueil-Malmaison) (Unknown); Nantes University Hospital (Other); Mental Health Center MGEN (Lille) (Unknown)
Responsible Party: Principal Investigator, Nicolas FRANCK, Pr, University professor - Hospital practitioner, Hôpital le Vinatier
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-A01676-37
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Chronic Schizophrenia
Keywords: Schizophrenia; Cognitive Remediation; Working abilities and social functioning
MeSH Terms: conditions — Schizophrenia; Social Adjustment | interventions — Cognitive Remediation; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RECOS (Experimental): The RECOS program (COgnitive REmediation for Schizophrenia) was designed by SBT Company and adapted by Vianin et al (2007) for specific use in schizophrenia. It includes computer based and paper and pencil exercises that target 6 main cognitive functions (selective attention; verbal memory; visuo-spatiale attention and memory, working memory, reasoning, and speed of execution) which have been recommended by the MATRICS consensus. Each exercise has 10 difficulty levels. Allocation of the training modules in RECOS is determined according to the standard scores obtained in the comprehensive neuropsychological assessment. Each patient participates in the module corresponding to his/her most altered cognitive area.
  Interventions: Behavioral: RECOS (COgnitive REmediation for Schizophrenia)
- TAU (Treatment as Usual) (Active Comparator): The treatment of the group TAU (Treatment As Usual) will consist of the usual care proposed by every service of the various inquiring centers involved. No additional session will be proposed.
  Interventions: Behavioral: TAU (Treatment As Usual)

INTERVENTIONS:
Behavioral: RECOS (COgnitive REmediation for Schizophrenia) — Every RECOS patient will benefit, with his therapist, from 2 sessions of 1 hour of training per week over a 14 weeks period (M1 to M3), plus 1 hour per week of task to be realized at home. All in all, it is thus about a training period of 42 hours.
  After remediation, the follow-up of the patient will be led by his therapist with monthly appointments during 6 months (M4 to M9).
  In parallel, neuropsychological and clinical scores will be assessed before (M0) and after the training period (M3), as well as at the end of the study (M9). Working and relational abilities will be assessed at the beginning and at the end of the working period (M4 and M9).
  Arms: RECOS
Behavioral: TAU (Treatment As Usual) — The treatment of the group TAU (Treatment As Usual) will consist of the usual care proposed by every service of the various inquiring centers involved. No additional session will be proposed.
  In parallel, neuropsychological and clinical scores will be assessed before (M0) and after the training period (M3), as well as at the end of the study (M9). Working and relational abilities will be assessed at the beginning and at the end of the working period (M4 and M9).
  Arms: TAU (Treatment as Usual)

SUMMARY:
This study, driven on schizophrenic patients, is aimed at :

1. Measuring the efficiency of the cognitive remediation program RECOS (COgnitive REmediation in Schizophrenia) on the capacity of the patients suffering from schizophrenia to improve the integration in sheltered employment (ESAT and EA).
2. Comparing the efficiency of the program of cognitive remediation RECOS (RECOS arm) to the one of an usual program of coverage/care (TAU arm = Treatment As Usual) on integration in sheltered employment of patients suffering from schizophrenia.
3. Realizing a comparative analysis, in both arms, of :

   1. the number of working hours achieved in sheltered environment during the 6 months following the two programs (reported to the working time planned by the contract of employment)
   2. the duration of such employments in sheltered areas.
4. Estimating the impact of RECOS on the neuropsychological variables, the symptomatology, the consciousness of the disorders(insight), the quality of life and the social autonomy before the treatment (month M0), at the end of the treatment (month M3), and 6 months later (month M9), and looking for a correlation between the improvement of these parameters and sheltered employment.
5. Estimating the impact of cognitive remediation on integration in sheltered employment.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 50 years.
* Schizophrenia according to the criteria of the DSM-IV-TR.
* Project of entry to ESAT or to EA in the 6 weeks which follow.
* IQ > 70 (F-NART).
* Stable symptomatology during the month preceding the inclusion.
* Psychotropic treatment unchanged during the month preceding the inclusion (change no more than 25 % posology).
* Overdrawn performances in at least one of the 6 functions estimated by the kit of neuropsychological tests.
* French mother tongue.
* Informed and signed consent by the patient.
* Agreement of the guardian (for protected adults).
* Membership in a national insurance scheme.

Exclusion Criteria:

* Dependence and recent abuses of cannabis (> 2 / week) or in any other substance (according to the criteria of the DSM-IV-TR), except tobacco.
* Neurological disorders of vascular, infectious or neurodegenerative origin; dyschromatopsie.
* Taking of medicine with somatic tropism having a cerebral or psychic impact (eg: corticoids).
* Simultaneous participation to any other program of remediation targeting the neurocognitive deficits.
* Resistance to neuroleptic.
* Reading and writing not acquired.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Number of worked hours during the first 6 months of the contract of employment | Outcome measures are daily assessed during 6 months (M4 to M9)
  Compared evolution in both arms (RECOS and TAU) of the number of worked hours, with regard to the number of hours planned in the contract of employment, during the 6 months following the entry in sheltered working environment (i.e. an external, validated and strong measure of the capacity of the patient to fit professionally).

SECONDARY OUTCOMES:
Compared evolution of the neuropsychological and clinical balance sheets between the beginning and the end of the Cognitive Remediation period (or the end of the "Treatment As Usual" period for the TAU arm) | Scores are assessed 3 times: at M0 (Inclusion), at M3 (after Cognitive Remediation or Treatment As Usual), and at M9 (6 month after end of treatment).
  Compared evolution, in both arms (RECOS and TAU) of the scores obtained in the different neuropsychological tests, and in the scales of clinical symptomatology (PANSS, questionnaires of insight, self-respect, well being, social autonomy, and cognitive complaint) at the moment of the inclusion (month M0), early after the training period of Cognitive Remediation or Treatment as Usual (M3), and 6 month after (M9).
Compared evolution of the neuropsychological and clinical balance sheets during the 6 first months of working contract (i.e. following the end of the training Cognitive Remediation period or after the "Treatment As Usual" period for the TAU arm). | Neuropsychological and clinical scores are assessed twice : at M3 (after Cognitive Remediation or Treatment As Usual), and at M9 (after 6 months of working period). Occupational integration (EATR) is assessed twice at the same moments (M3 & M9).
  Compared evolution, in both arms (RECOS and TAU) of the scores obtained in the different neuropsychological tests, and in the scales of occupational integration (EATR), clinical symptomatology (PANSS, questionnaires of insight, self-respect, well being, social autonomy, and cognitive complaint) after the training period of Remediation and at the moment of the entry in sheltered working environment (month M3), and 6 months later (month M9).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas FRANCK, Professor, Principal Investigator — University Service of Rehabilitation (SUR) of the Vinatier Hospital; Brice MARTIN, Doctor, Study Director — University Service of Rehabilitation (SUR) of the Vinatier Hospital; Isabelle AMADO, Doctor, Study Director — Center of Study and Clinical Research (CERC) of the Ste Anne Hospital; Corinne LAUNAY, Doctor, Study Director — Center of Study and Clinical Research (CERC) of the Ste Anne Hospital; Marie-Cécile BRALET, Doctor, Study Director — Service CRISALID of the Clermont-de-l'Oise's Hospital; Elisabeth GIRAUD-BARO, Doctor, Study Director — Saint-Egrève's Hospital; Julien DUBREUCQ, Doctor, Study Director — Saint-Egrève's Hospital; Pascal BLOCH, Doctor, Study Director — Niort's Hopsital; Christophe LANCON, Professor, Study Director — Sainte Marguerite Hospital; Eric FAKRA, Doctor, Study Director — Sainte Marguerite Hospital; Jean-Michel ZAKOIAN, Professor, Study Chair — Ecole Nationale de la statistique; Christian FRANCQ, Professor, Study Chair — Ecole Nationale de la statistique; Pascal VIANIN, Doctor, Study Chair — Centre Hospitalier Universitaire Vaudois; Nathalie GUILLARD-BOUHET, Doctor, Study Director — Henri Laborit Hospital; Muriel BONAÏTI, Doctor, Study Director — Saint Cyr Hospital; Jérome GRAUX, Doctor, Study Director — Tours University Hospital; Bernard DUBOUIS, Doctor, Study Director — Mental Health Center MGEN (Rueil-Malmaison); Vincent SCHAER, Doctor, Study Director — Mental Health Center MGEN (Rueil-Malmaison); Jérome SETTON, Doctor, Study Director — Mental Health Center MGEN (Rueil-Malmaison); Vincent DELAUNAY, Doctor, Study Director — Nantes University Hospital; Marion CHIRIO-ESPITALIER, Doctor, Study Director — Nantes University Hospital; Ingrid DUR, Doctor, Study Director — Mental Health Center MGEN (Lille); Sophie DELILLE, Doctor, Study Director — Mental Health Center MGEN (Lille); Olivier MAZAS, Doctor, Study Director — Mental Health Center MGEN (Lille)
Locations (13):
- France (13):
  - Hôpital Le Vinatier Pôle Centre, Bron
  - Hôpital Le Vinatier Pôle Est, Bron
  - Mental Health Center (MGEN), Lille
  - Hôpital Ste Marguerite, Marseille
  - Nantes University Hospital, Nantes
  - Centre Hospitalier de Niort, Niort
  - Hôpital Ste Anne, Paris
  - Centre Hospitalier Henri Laborit, Poitiers
  - Mental Health Center (MGEN), Rueil-Malmaison
  - Saint-Cyr Hospital, Saint-Cyr-au-Mont-d'Or
  - Centre Hospitalier de St-Egrève, Saint-Egrève
  - Centre de Santé Mentale Angevin (CESAME), Sainte-Gemmes-sur-Loire
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deppen P, Sarrasin Bruchez P, Dukes R, Pellanda V, Vianin P. [Cognitive remediation program for individuals living with schizophrenia (Recos): preliminary results]. Encephale. 2011 Sep;37(4):314-21. doi: 10.1016/j.encep.2011.02.002. Epub 2011 Apr 9. French. PMID 21981893
- [Background] Franck N, Duboc C, Sundby C, Amado I, Wykes T, Demily C, Launay C, Le Roy V, Bloch P, Willard D, Todd A, Petitjean F, Foullu S, Briant P, Grillon ML, Deppen P, Verdoux H, Bralet MC, Januel D, Riche B, Roy P; Other members of the Cognitive Remediation Network; Vianin P. Specific vs general cognitive remediation for executive functioning in schizophrenia: a multicenter randomized trial. Schizophr Res. 2013 Jun;147(1):68-74. doi: 10.1016/j.schres.2013.03.009. Epub 2013 Apr 9. PMID 23583327